CLINICAL TRIAL: NCT06456684
Title: AV133 Longitudinal Imaging Study in Patients With Early and Prodromal Parkinson's Disease
Brief Title: AV133 Longitudinal Imaging Study in Patients With Early and Prdromal Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The Michael J. Fox Foundation for Parkinson's Research (Unknown); XINGIMAGING LLC (Unknown); Naming MITRO Pharmaceutical Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: 114
Record Dates: First submitted 2024-03-04; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: PD; [18F]promethazine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early-stage Parkinson's disease
  Interventions: Diagnostic Test: Fluoro[18F]promethazine
- prodromal Parkinson's disease
  Interventions: Diagnostic Test: Fluoro[18F]promethazine

INTERVENTIONS:
Diagnostic Test: Fluoro[18F]promethazine — It is the first F-18-labeled VMAT2 imaging agent for PET imaging that is currently being used in the clinic internationally. In the brains of Parkinson's disease (PD) patients, the target binding of fluoro[18F]promethazine was significantly reduced compared with that of normal controls, with an 81% reduction in the posterior region of the nucleus accumbens, a 70% reduction in the anterior region of the nucleus accumbens, and a 48% reduction in the caudate nucleus; the radioactivity uptake in the caudate nucleus of PD patients was correlated with the extent of their disease

SUMMARY:
A total of 38 patients with early-stage Parkinson's disease and 38 patients with prodromal Parkinson's disease are planned to be enrolled in this study and examined for longitudinal changes in [18F]AV-133 through follow-up, thereby informing the design of future therapeutic trials utilizing [18F]AV-133 as a marker of disease progression.

DETAILED DESCRIPTION:
This study is a longitudinal study designed to assess the progression of [18F]AV-133 imaging in patients with prodromal and early stages of Parkinson's disease . Approximately 38 patients with early PD and 38 subjects in the prodromal phase will be enrolled in the study. All subjects will undergo imaging assessment with [18F]AV-133 at baseline and every 12 months thereafter, clinical (motor, neuropsychiatric and cognitive) assessment, and biospecimen collection for bioanalysis. The study duration for each subject will be approximately 27 months, including a 60-day screening period and a 24-month follow-up assessment period. Data collection will be performed uniformly for all participants according to the protocol developed.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Parkinson's disease： Men or women aged 30 years or older at the time of diagnosis of Parkinson's disease.

Patients must have at least two of the following: resting tremor, bradykinesia, tonicity (must have resting tremor or bradykinesia); or asymmetric resting tremor or asymmetric bradykinesia.

Time to diagnosis of Parkinson's disease at screening was 2 years or less. Hoehn & Yahr staging stage I or II at baseline. AV133 PET scan suggestive of vesicular monoamine transporter 2 (VMAT2) deficiency.

Able to provide informed consent. Not yet started on PD medication.

Clinical diagnosis of Parkinson's disease in the prodromal phase： Subjects confirmed eligible based on existing predictive criteria Olfactory dysfunction confirmed by olfactory testing. Other predictive criteria based on general risk, such as first-degree biological relatives, known Parkinson's disease risk including RBD, or known genetic variants associated with Parkinson's disease risk (LRRK2 or GBA).

Men or women 60 years or older (or 30 years or older for subjects with SNCA or rare genetic variants such as Parkin or Pink1) AV133 deficiency as determined by visual assessment (screening PET scan) Subjects taking any of the following medications: α-methyldopa, methylphenidate, amphetamine derivatives, or modafinil must be willing and medically able to discontinue the medication for at least 5 half-lives prior to PET imaging.

Able to provide informed consent. Not yet started on PD medication.

Exclusion Criteria：

Currently taking levodopa, dopamine agonists, MAO-B inhibitors, amantadine, or other anti-Parkinson's disease medications.

Diagnosed with dementia and related cognitive impairment disorders. Received any of the following medications that may interfere with PET imaging of the dopamine transporter protein within 1 month prior to screening: antipsychotics, metoclopramide, α-methyldopa, methylphenidate, reserpine, modafinil, or amphetamine derivatives.

Current clinically significant cardiovascular disease or screening ECG abnormalities (including but not limited to QTc > 450 ms) Currently taking medications known to cause QT prolongation; Use of an investigational drug or device within 60 days prior to baseline (dietary supplements taken outside of a clinical trial are not exclusionary, e.g., coenzyme Q10).

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 38 patients with early-stage Parkinson's disease and 38 patients with prodromal Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
to assess the mean rate of change and variability of AV133 imaging results | baseline the 12 months and 24 months
  to assess the mean rate of change and variability of AV133 imaging results from baseline at 12 and 24 months follow-up in patients with prodromal and

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No